CLINICAL TRIAL: NCT06375993
Title: A Phase 1 Study of ADI-001 Anti-CD20 CAR-engineered Allogeneic Gamma-Delta (γδ) T Cells in Adults With Autoimmune Disease
Brief Title: A Phase 1 Study of ADI-001 in Autoimmune Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Adicet Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ADI-202300103
Record Dates: First submitted 2024-04-17; First posted 2024-04-19 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-01

CONDITIONS: Lupus Nephritis; Autoimmune Diseases; Systemic Sclerosis (SSc); Systemic Lupus Erythematosus (SLE); ANCA-Associated Vasculitis (AAV); Idiopathic Inflammatory Myopathies; Stiff Person Syndrome
MeSH Terms: conditions — Lupus Nephritis; Autoimmune Diseases; Scleroderma, Systemic; Lupus Erythematosus, Systemic; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Myositis; Stiff-Person Syndrome | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: 3+3 Dose Escalation Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- ADI-001 Dose Escalation (Experimental): ADI-001 is administered via infusion with ascending dose levels as a single dose to determine the maximum tolerated dose (MTD) or maximum assessed dose (MAD) of ADI-001.
  Interventions: Drug: ADI-001; Drug: Fludarabine; Drug: Cyclophosphamide
- ADI-001 Dose Extension (Experimental): After dose level has been declared safe, additional patients can be enrolled at the declared safe dose to further investigate the safety profile of ADI-001.
  Interventions: Drug: ADI-001; Drug: Fludarabine; Drug: Cyclophosphamide
- ADI-001 Dose Expansion (Experimental): Dose Expansion ADI-001 is administered via infusion at the MTD/MAD to confirm recommended phase 2 dose (Part 2).
  Interventions: Drug: ADI-001; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: ADI-001 — Anti-CD20 CAR-T
Drug: Fludarabine — Chemotherapy for Lymphodepletion
Drug: Cyclophosphamide — Chemotherapy for Lymphodepletion

SUMMARY:
ADI-202300103 is a phase 1 multicenter, open label, dose finding and dose expansion, safety/efficacy study in patients with autoimmune disease. The study will consist of different periods including screening, lymphodepletion, treatment, and follow-up

ELIGIBILITY:
Inclusion Criteria:

For Cohort 1: Subjects with LN:

1. Clinical diagnosis of systemic lupus erythematosus (SLE) per 2019 European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) classification criteria (Aringer 2019)
2. Active kidney disease with biopsy-proven active LN Class III or IV (coexistent class V permitted) (per 2018 International Society of Nephrology [ISN]/Renal Pathology Society [RPS] criteria); biopsy should be performed within 6 months before enrolling in the study
3. ECOG performance ≤ 2
4. Proteinuria (or urine protein creatinine ratio [UPCR]) > 1g / 24 hours

For Cohort 1: Subjects with SLE with Extrarenal Involvement

1. Clinical diagnosis of systemic lupus erythematosus (SLE) per 2019 European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) classification criteria (Aringer 2019).
2. Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score ≥ 8 with a clinical SLEDAI-2K score (SLEDAI-2K not including points for anti-dsDNA and/or low complement) ≥ 6 and/or ≥ 1 British Isles Lupus Assessment Group (BILAG)-2004 Category A
3. Positive anti-nuclear antibody (ANA) test results and/or a positive anti-dsDNA and/or anti-Smith antibodies above the ULN
4. Estimated creatinine clearance ≥ 60 mL/min
5. Inadequate response in terms of active disease despite treatment with current standard of care for SLE including corticosteroids and at least 2 SLE therapy

For Cohort 2: Subjects with SSc

1. Disease duration ≤ 6 years (from onset of first non-Raynaud manifestation)
2. Participants with diffuse cutaneous SSc with worsening skin disease, must meet both of the following criteria: mRSS ≥ 15 at screening AND one of the following within 6 months prior to screening: (i) mRSS increase of ≥ 3 units in the total mRSS, OR (ii) Involvement of 1 new body area, OR (iii) Increase in mRSS ≥ 2 units in 1 body area
3. Participants with diffuse or limited cutaneous SSc and ILD must meet both of the following criteria: ILD, i.e. fibrosis on HRCT within 4 months of screening AND Progression of ILD by FVC or HRCT in previous 24 months
4. FVC ≥ 45% predicted, DLCO ≥ 40%
5. Exclude PAH defined as RVSP ≥ 45 mmHg or right atrial or ventricular enlargement or dilatation, or renal crisis within 1 year of enrollment

For Cohort 3: Subjects with AAV

1. Diagnosis of AAV defined as either GPA or MPA according to the 2012 Chapel Hill Consensus Conference
2. Positive for PR3-ANCA or MPO-ANCA
3. Relapsed or refractory AAV after at least 1 standard-of-care immunosuppressive regimen in addition to steroids.
4. Severe disease (i.e., presence of one or more major AAV sign or symptom per the BVAS or ≥ 3 minor items, or at least the 2 renal items of proteinuria and hematuria due to vasculitis)
5. Adequate renal function: CrCl ≥ 30 mL/min
6. Proteinuria ≤ 8 g/24 hour

For Cohort 4: Subjects with Idiopathic Inflammatory Myopathies

1. Meets the 2017 ACR/EULAR classification criteria (Lundberg 2017) for probable/definite IIM
2. Muscle weakness defined as Manual Muscle Testing (MMT)-8 score < 142/150, and ≥ 2 of the following abnormal core set measures: (i) Patient global assessment VAS ≥ 2 cm (on 10-cm VAS), (ii) Physician global assessment VAS ≥ 2 cm (10-cm VAS), (iii) HAQ-DI > 0.25 , (iv) Extra-muscular global activity VAS ≥ 2 cm (10-cm VAS)
3. Active disease defined as ≥ 1 of the following signs in the past 4 months: a) Elevated serum CK or aldolase levels ≥ 3 times ULN; b) Active myositis by muscle biopsy, muscle MRI, or EMG; c) Active DM rash and CDASI >14; d) Active interstitial lung disease
4. Positivity for ≥ 1 myositis-specific antibody or myositis-associated antibody at screening
5. Inadequate response or intolerance/contraindication to glucocorticoids and to ≥ 2 immunosuppressants for 3 months/drug

For Cohort 4: Subjects with Stiff Person Syndrome

1. Meets the 2009 criteria for diagnosis of stiff person syndrome (SPS) (Dalakas 2009): (a) Stiffness of the axial muscles, particularly the abdominal and thoraco-lumbar paraspinals, leading to hyperlordosis; (b) Superimposed painful spasms triggered by unexpected tactile or auditory stimuli; (c) Severe anxiety with task-specific phobias especially in anticipation of physically challenging tasks; (d) Electromyographic evidence of continuous motor unit activity of agonist and antagonist muscles; (e) Absence of other neurological findings that may suggest an alternative diagnosis; (f) Highly positive anti-GAD titer (> 10,000 IU/mL in serum by ELISA or detectable in CSF)
2. Inadequate response or intolerance or contraindication to ≥ 1 treatment including chronic IVIG or other biologic

Exclusion Criteria:

For all Subjects:

1. Presence of severe liver disease, Child-Pugh class B or C.
2. Prior treatment with any gene therapy, genetically modified cell therapy, or adoptive T cell therapy.
3. Autoimmune disease requiring prednisone higher than 0.5 mg/kg/day (or corticosteroid equivalent).
4. Subjects unwilling to participate in an extended safety monitoring period (LTFU protocol)
5. History of a clinically significant infection (including sepsis, pneumonia, bacteremia, fungal, viral and opportunistic infections) within 4 weeks prior to first dose of study drug which in the opinion of the Investigator may compromise the safety of the subject in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-11-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The Incidence of Subjects with Dose Limiting Toxicities within each dose level cohort | 28 Days
  This primary endpoint will be used to determine the Maximum Tolerated Dose (MTD) or Maximum Assessed dose (MAD)
Proportion of treatment emergent and treatment related adverse events | 2 year
  This primary endpoint will be used to determine the MTD/MAD of ADI-001

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Adicet Clinical Trials, Redwood City, California
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York

IPD SHARING:
Plan to Share IPD: No